CLINICAL TRIAL: NCT05117983
Title: Non-invasive Brain Stimulation Normalizes Dopaminergic Transmission in the Frontostriatal Circuit to Alleviate Depression With Metabolic Disorders.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-110-005
Record Dates: First submitted 2021-09-28; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: Depression
Keywords: Depression; Dopamine (DA); Frontostriatal (FS) circuit; Metabolic disorder; Repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Depression; Metabolic Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDD patient with HRSD score of at least 18 (Active Comparator): MDD patients who meet the DSM-5 diagnostic criteria of MDD and their current episode show a Hamilton Rating Scale for Depression (HRSD) score of at least 18
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- BD patient with HRSD score of at least 18 (Active Comparator): BD patients who meet the DSM-5 diagnostic criteria of BD and their current depression episode show a Hamilton Rating Scale for Depression (HRSD) score of at least 18
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — Real-time MRI-guided neuronavigation with a Visor neuronavigation system (ANT Neuro, Enschede, Netherlands) will be used for coil positioning. Left dorsolateral prefrontal cortex target is located in each participant.
  Other Names: Antidepressants

SUMMARY:
Depression and metabolic disorder (MetD) are two of the most common and debilitating disorders worldwide, occurring with significant rates of comorbidity. This is a major clinical challenge as the outcomes of both conditions are worsened. Studies have uncovered that depression and metabolic disorder are associated with chronic, low-grade inflammation. In brain circuit level, patients with depression are characterized with aberrant frontostriatal (FS) circuit connectivity and reduced activity level that also associated with metabolic comorbidity. In neurotransmitter level, the dopaminergic pathway, that could be feedback regulated by immune and metabolic factors, has long been known to involve in emotional and metabolic homeostasis. More importantly, this dopamine (DA) input is critical to shaping the FS circuit-level dynamic connectivity and plasticity. Therefore, this study hypothesizes that inflammatory and metabolic dysregulations on DA transmission link to the aberrant FS function that cause mood and metabolic syndromes. To clarify the underlying mechanisms, 90 patients who meet the DSM-5 diagnostic criteria of major depressive episode in either major depressive disorder or bipolar disorder are planned to be recruit. FS functional connectivity and activation, before and after receiving 10 Hz repetitive transcranial magnetic stimulation (rTMS) to left dorsolateral prefrontal cortex will be measured. Then systemically analyze participants' clinical symptomology, neurocognitive function, inflammation and metabolic status. Possible correlations between indices, the effects of rTMS and differences between groups will be tested. Results could provide a chance for further understanding the pathophysiology of depression with MetD and comparing between unipolar and bipolar depression, and developing brain circuit based non-invasive brain stimulation personalized treatment for depression with MetD to achieve a better outcome.

DETAILED DESCRIPTION:
Depression and metabolic disorder (MetD) are two of the most common and debilitating disorders worldwide, occurring with significant rates of comorbidity. This is a major clinical challenge as the outcomes of both conditions are worsened. Studies have uncovered that depression and metabolic disorder are associated with chronic, low-grade inflammation. In brain circuit level, patients with depression are characterized with aberrant frontostriatal (FS) circuit connectivity and reduced activity level that also associated with metabolic comorbidity. BD patients also showed functional anomalies in the VS and FS circuits with reduced neural flexibility of hedonic signaling in response to stress. The dysfunctional FS circuits also link to the metabolic comorbidities in patients with mood disorders. Regarding metabolic control, the FS functional connectivity changes affect food craving. And the altered reciprocal loop from the medial prefrontal cortex could regulate eating behavior and metabolic disturbance. In neurotransmitter level, the dopaminergic pathway, that could be feedback regulated by immune and metabolic factors, has long been known to involve in emotional and metabolic homeostasis. More importantly, this dopamine (DA) input is critical to shaping the FS circuit-level dynamic connectivity and plasticity. Disruptions in the dopamine (DA) system have been observed in psychiatric disorders. MDD might involve DA reductions that could result from either diminished DA release from presynaptic neurons or impaired signal transduction, either due to changes in receptor number or function and/or altered intracellular signal processing. Therefore this study hypothesizes that inflammatory and metabolic dysregulations on DA transmission link to the aberrant FS function that cause depression and MetD. To clarify the underlying mechanisms, unipolar and bipolar depression patients will be enrolled to measure the FS functional connectivity and activation, before and after receiving 10 Hz repetitive transcranial magnetic stimulation (rTMS) to left dorsolateral prefrontal cortex. Then systemically analyze participants' clinical symptomology, neurocognitive function, inflammation and metabolic status. Possible correlations between indices, the effects of rTMS and the possible differences between unipolar and bipolar depression patients will be tested. Results could provide a chance for further understanding the pathophysiology and better treatment of depression with MetD, finding biomarkers for subgrouping depression between unipolar depression and bipolar depression, predicting outcomes to brain circuit based personalized rTMS treatment for depression with MetD.

The specific aims of the project are:

Aim 1: To find the biological homogeneousness among depression with MetD by investigate the associations between (1) FS circuit connectivity and clinical (mood and metabolic) symptoms, and (2) FS circuit activation and clinical (mood and metabolic) symptoms in both unipolar and bipolar depressed individuals.

Aim 2: To confirm the role of FS in depression with MetD by applying rTMS to test its effects on (1) clinical symptoms, (2) FS circuit activation, (3) FS circuit connectivity and (4) find predictors for the rTMS treatment response.

Aim 3: To study the bidirectional inflammatory and metabolic feedback regulations of the DA transmission in FS circuit in depression with MetD by investigate the associations between (1) FS circuit activation, and (2) FS circuit connectivity and systemic inflammatory/ metabolic regulators both before and after rTMS treatments.

ELIGIBILITY:
Inclusion Criteria:

* (1)Signed informed consent by patient or legal representative;
* (2) male or female patient aged ≧20 and ≦70 years;
* (3) a diagnosis of MDD or BD according to DSM criteria made by a specialist in psychiatry;
* (4) a total score of at least 18 in the Hamilton Rating Scale for Depression (HDRS) at the screening stage;
* (5) patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

* (1) women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study;
* (2) females who are pregnant or breast-feeding;
* (3) other major DSM 5 diagnoses other than mood disorders, except for tobacco use disorder and anxiety disorder;
* (4) current evidence of an uncontrolled and/or clinically significant medical condition, e.g. patients with extensive area of ischemic bruise, multiple sclerosis, cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation;
* (5) history of seizure or epilepsy;
* (6) history of neurological diseases or traumatic brain injury;
* (7) history of brain lesion, having received neurosurgery, meningitis or encephalitis;
* (8) exacerbation of symptom severity, presenting severe suicidal ideation or self harm behavior during the screen or study period;
* (9) presence of devices, e.g. pacemakers, cochlear prosthesis, neuro-stimulators, magnetic cochlear prosthesis, intracranial/intraocular metallic fragments;
* (10) patient has received electroconvulsive therapy (ECT) within 3 months prior to the first intervention of the treatment;
* (11) skin lesion at local site receiving rTMS stimulation;
* (12) those who cannot tolerate the side effects or ever developed sleep disorder while receiving rTMS therapy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline mood symptom severity at several timepoints over 3 months | Week 0, Week 1, Week 2, Week 3, Week 4, Week 8, Week 12.
  Evaluation for disease severity by using the Hamilton Rating Scale for Depression (HAM-D) by trained senior psychiatrists. The same rater administers the scale for each patient.
Iowa gambling task (IGT) with functional MR imaging | Week 0
  The subject will be asked to turn a card from 4-decks voluntarily, and maximize gains and minimize losses during the game.
Change from baseline functional connectivity maps at 3 months | Week 0, Week 12
  A 2-sample independent t-test will be employed to analyze the functional connectivity maps using SPM 12. Statistical maps will be computed to identify changes in striatum-seeded functional connectivity for between-group comparisons. The age will be regressed out as a covariate of non-interest. Significance will be threshold at the uncorrected voxel level p=0.001, followed by the FWE- corrected cluster level p=0.05.
Change from baseline homeostasis model assessment-estimated insulin resistance (HOMA-IR) index at several timepoints within 3 months | Week 0, Week 4, Week 8, Week 12
  The homeostasis model assessment-estimated insulin resistance (HOMA-IR) index is calculated as the product of the fasting plasma insulin level (uIn/ml) and the fasting plasma glucose level (mg/dl), divided by 405. Insulin resistance is defined as HOMA-IR ≥2.5.
Change from baseline body mass index (BMI) at several timepoints within 3 months | Week 0, Week 4, Week 8, Week 12
  Body weight (to the nearest 0.1 kg), body height (to the nearest 0.1 cm) will be measured and BMI (kg/m2) will be calculated accordingly.
Change from baseline waist and hip circumference at several timepoints within 3 months | Week 0, Week 4, Week 8, Week 12
  Waist and hip circumference (to the nearest 0.1 cm) will be measured.
Change from baseline fasting serum leptin level at several timepoints within 3 months | Week 0, Week 4, Week 8, Week 12
  Measured using ELISA method (Linco Research, USA). The limit of detection was 0.5 ng/mL, and the intra- and interassay coefficients of variation were 7% and 9%, respectively.
Change from baseline fasting serum lipid level at several timepoints within 3 months | Week 0, Week 4, Week 8, Week 12
  Fasting total cholesterol, high density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL) and triglyceride (TG) concentrations will be measured.
Change from baseline immunological markers at several timepoints within 3 months | Week 0, Week 2, Week 3, Week 4, Week 8, Week 12
  The fasting plasma CRP level will be assessed using an high-sensitivity CRP ELISA kit (Bender MedSystems, USA), for which the limit of detection was 3 pg/mL and the intra- and inter-assay coefficients of variation were 6.9% and 13.1%, respectively. The other immunological parameters to be analyzed include TNF-α, TGF-β1, IL-1, IL-8 and IL-10.
Change from baseline neurocognitive performance at 3 months | Week 0, Week 12
  Neurocognitive performance will be assessed using Continuous Performance Test (CPT), Finger-Tapping Test (FTT) and Wisconsin Card-Sorting Test (WCST).
Change from baseline social cognitive function at 3 months | Week 0, Week 12
  Mayer-Salovey-Caruso emotional Intelligent Test (MSCEIT): four branches: perceiving emotion (consisting of two tasks: face and picture tasks), facilitating emotion, understanding emotion, and managing emotion (Mayer, Salovey, Caruso, & Sitarenios, 2003). The results will be scaled to a standard score based on the weight from the representative adult population (regarding age, gender, and ethnicity) in an extremely large sample of people (5,000). The reliability and validity of MSCEIT V2.0 have been proved before.
Change from baseline autonomic nervous system performance at several timepoints within 3 months | Week 0, Week 4, Week 12
  Cardiac autonomic function will be calculated by the geometric method, which is based on short-term measurements of the interbeat interval (IBI) [82]. Power spectral density analysis of HRV will be performed by fast Fourier transformation [83].

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan